CLINICAL TRIAL: NCT06547632
Title: ClearPetra™ Vacuum-assisted Ureteral Access Sheath vs Traditional Approach in Retrograde Intrarenal Surgery. A Randomized Controlled Trial
Brief Title: ClearPetra™ Vacuum-assisted Ureteral Access Sheath vs Traditional Approach
Acronym: VA-UAS vs trad
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Wilson Molina, Professor of Urology, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00161273
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Nephrolithiasis; Kidney Stone
Keywords: Nephrolithiasis; Kidney Stone; ClearPetra; Ureteral access sheath
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 1. RIRS WITH VACUUM-ASSISTED URETERAL ACCESS SHEATH (Active Comparator): In Arm 1, participants will undergo RIRS with ClearPetra™ vacuum-assisted ureteral access sheath.
  Participants will undergo RIRS per standard of care.
  Interventions: Device: ClearPetra Ureteral access sheath
- 2. RIRS WITH TRADITIONAL APPROACH (No Intervention): In Arm 2, participants will undergo RIRS a traditional approach (no sheath or non-vacuum-assisted sheath). The treating investigator will decide whether to use a regular UAS based on their preference and/or availability.
  * No ureteral access sheath
  * Navigator™ Ureteral Access Sheath 11/13 Fr (Boston Scientific®)
  * Navigator™ Ureteral Access Sheath 12/14 Fr (Boston Scientific®)

INTERVENTIONS:
Device: ClearPetra Ureteral access sheath — Patients will be randomly assigned (1:1) to vacuum-assisted (ClearPetra) or traditional approach group for retrograde intrarenal surgery according to standard of care.
  Arms: 1. RIRS WITH VACUUM-ASSISTED URETERAL ACCESS SHEATH

SUMMARY:
Ureteroscopy has been considered the best approach when treating renal stones smaller than 2 cm. This procedure is usually performed together with ureteral access sheaths, which helps protect the ureter mucosa and lowers intrarenal pressure.

Recently, a new vacuum-assisted ureteral access sheath called ClearPetra has entered US market and allows for continuous stone fragmentation and aspiration.

Because there is little information on comparing this device with traditional approach (no sheath or non-vacuum-assisted sheath) in American population, we aim to compare those devices in terms of their ability to clear the kidney from kidney stones, as well as reduce infection rates postoperatively.

DETAILED DESCRIPTION:
Retrograde intrarenal surgery (RIRS) is now considered gold-standard for treatment of renal stones smaller than 2 cm. This procedure often employs a ureteral access sheath (UAS), as it helps to reduce intrarenal pressure and protects the ureter mucosa when basketing is required. However, the challenge imposed by residual stone fragments and sepsis remains. Additionally, natural elimination of residual stone fragments may induce renal colic, hematuria an even the potential for new stone development. Recently, a new vacuum-assisted ureteral access sheath (VA-UAS) named ClearPetra™ provides concomitant stone fragmentation and aspiration.

The new ClearPetra™ vacuum assisted ureteral access sheath allows simultaneous fragmentation and extraction of stones. It is a disposable access sheath equipped with a continuous flow aspiration mechanism. Previous studies have demonstrated the safety and effectiveness of ClearPetra™ in RIRS Comprehensive comparative investigations between ClearPetra™ and traditional UAS in RIRS are lacking in American population. We aim to compare the outcomes of using VA-UAS (ClearPetra™) or traditional approach (no sheath or non-vacuum-assisted sheath) to treat patients with stone burden between 1.0 - 2.5 cm.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females over18 years of age
2. Undergoing primary flexible ureteroscopy for retrograde intrarenal surgery
3. Total stone burden between 1.0 to 2.5 cm

Exclusion Criteria:

1. Undergoing bilateral stone treatment during the same procedure
2. Patients with known genitourinary anatomical abnormalities
3. Uncorrected coagulopathy
4. Patients with urinary diversions
5. Chronic external urinary catheters
6. Women who are pregnant
7. Immunosuppressed patients
8. Non-elective procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Stone Free Status between ClearPetra and traditional approach | 90 days
  Stone free is defined as no residual stones >2mm in post operative CT scan

SECONDARY OUTCOMES:
Total operative time between ClearPetra and traditional approach | 1 day
  Time from scope insertion to scope removal from the patient
Urinary tract infection between ClearPetra and traditional approach | 30 days of procedure
  Data collection searching for urine tract infection signs, symptoms, antibiotic administration and culture

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Molina, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonyali S. Suctioning ureteral access sheath use in flexible ureteroscopy might decrease operation time and prevent infectious complications. World J Urol. 2019 Feb;37(2):393-394. doi: 10.1007/s00345-018-2510-5. Epub 2018 Sep 26. No abstract available. PMID 30259124
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART I. J Urol. 2016 Oct;196(4):1153-60. doi: 10.1016/j.juro.2016.05.090. Epub 2016 May 27. PMID 27238616
- [Background] Chen Y, Zheng L, Lin L, Li C, Gao L, Ke L, Kuang R, Chen J. A novel flexible vacuum-assisted ureteric access sheath in retrograde intrarenal surgery. BJU Int. 2022 Nov;130(5):586-588. doi: 10.1111/bju.15873. Epub 2022 Sep 6. No abstract available. PMID 35986898